CLINICAL TRIAL: NCT02414581
Title: Mouthwash With Chlorhexidine 0.12%/Ethyl Alcohol 7% Compared to Ethyl Alcohol 7% to Reduce the Rate Oral Colonization by Gram-negative Bacteria in Patients With Chemotherapy
Brief Title: Mouthwash With Chlorhexidine 0.12%/Ethyl Alcohol 7% Compared to Ethyl Alcohol 7%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Collaborators: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Lauro Fabian Amador Medina, Researcher, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ci-HRAEB-2015-004
Record Dates: First submitted 2015-04-03; First posted 2015-04-10 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2016-09

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Chlorhexidine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chlorhexidine 0.12% & Ethyl Alcohol 7% (Experimental): Chlorhexidine 0.12% and Ethyl Alcohol 7% mouthwashes 15ml by 30 seconds, twice day for 9 days.
  Interventions: Drug: chlorhexidine 0.12%/Ethyl alcohol 7%
- Ethyl Alcohol 7% (Active Comparator): Ethyl Alcohol 7% without chlorhexidine mouthwashes 15ml by 30 seconds, twice day for 9 days.
  Interventions: Drug: Ethyl Alcohol 7%
- Chlorhexidine 2% & Ethyl Alcohol 7% (Experimental): Chlorhexidine 2% and Ethyl Alcohol 7% mouthwashes 15ml by 30 seconds, once day for 3 days.
  Interventions: Drug: Chlorhexidine 2%/Ethyl alcohol 7%

INTERVENTIONS:
Drug: chlorhexidine 0.12%/Ethyl alcohol 7% — Mouth rinses with chlorhexidine 0.12%-based solution
  Arms: Chlorhexidine 0.12% & Ethyl Alcohol 7%
Drug: Ethyl Alcohol 7% — Mouth rinses with Ethyl Alcohol 7%-based solution
  Arms: Ethyl Alcohol 7%
Drug: Chlorhexidine 2%/Ethyl alcohol 7% — Mouth rinses with chlorhexidine 2%-based solution
  Arms: Chlorhexidine 2% & Ethyl Alcohol 7%

SUMMARY:
Clinical triple-blind randomized controlled trial to assess the use of two different mouthwashes to reduce the oral colonization by gramnegative bacteria in patients with chemotherapy

DETAILED DESCRIPTION:
Clinical triple-blind randomized controlled trial.

With two arms to the study:

1. Mouth rinses with chlorhexidine-based solution at a concentration of 0.12%, using as a vehicle to 7% ethyl alcohol.
2. Mouthwashes with solution based only 7% ethyl alcohol.

GOAL. Assess whether there decrease in the rate of oral colonization by gram-negative bacteria in patients with chemotherapy by using chlorhexidine mouthwash.

SPECIFIC OBJECTIVES:

1. The rate of the oral colonization by gram-negative bacteria initiation of chemotherapy.
2. The rate of oral colonization by gram-negative bacteria after 10 days of initiation of chemotherapy.
3. Identify microbiologically gram-negative bacteria colonizing the oral cavity.

SECONDARY OBJECTIVES

1. The presence of severe neutropenia and fever in each study group during the first 10 days of starting treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18years, no upper age limit.
2. Acceptance of participation in the study.
3. Signature of informed consent.
4. Inpatient and remain hospitalized for at least 10 days.
5. The following haematological diagnosis:

   1. acute lymphoblastic leukemia.
   2. acute myelogenous leukemia.
   3. relapsed non-Hodgkin lymphoma.
6. Receiving Chemotherapy scheme as a treatment for the underlying disease

Exclusion Criteria:

1. Patients who choose not to participate in the study.
2. Patients in whom no possible mouthwashes.
3. Patients who willingly choose to withdraw from the study.
4. Patients who develop conditions in which the administration is not possible rinses.
5. Duration of hospital stay less than 10 days, regardless of cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of oral colonization by gram-negative bacteria | 10 days

SECONDARY OUTCOMES:
Rate of oral colonization by gram-negative bacteria at the start of chemotherapy in each study arm. | Baseline
Identify microbiologically gram-negative bacteria that colonize the oral cavity in each study arm | 10 days
Number of participants with presence of severe neutropenia and fever in each study group. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Lauro F Amador, Researcher, Principal Investigator — Hospital Regional Alta Especialidad Bajio
Locations (1):
- Hospital Regional Alta Especialidad Bajio, León, Guanajuato, Mexico

REFERENCES:
- [Result] Pitten FA, Kiefer T, Buth C, Doelken G, Kramer A. Do cancer patients with chemotherapy-induced leukopenia benefit from an antiseptic chlorhexidine-based oral rinse? A double-blind, block-randomized, controlled study. J Hosp Infect. 2003 Apr;53(4):283-91. doi: 10.1053/jhin.2002.1391. PMID 12660125